CLINICAL TRIAL: NCT00179127
Title: Early Use of Insulin Glargine in Diabetic Ketoacidosis
Brief Title: Use of Insulin Glargine to Treat Diabetic Ketoacidosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 040643
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Results first posted 2018-07-16 (Actual); Last update posted 2018-07-16 (Actual); Status verified 2018-06

CONDITIONS: Diabetic Ketoacidosis
Keywords: Pediatrics; Diabetes; Emergency Care; Endocrinology; Critical Care
MeSH Terms: conditions — Diabetic Ketoacidosis; Diabetes Mellitus | interventions — Insulin Glargine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glargine (Experimental): 0.3u/kg of glargine, subcutaneously, once
  Interventions: Drug: glargine
- Placebo (Placebo Comparator): 0.3u/kg of saline, subcutaneously, once
  Interventions: Drug: saline

INTERVENTIONS:
Drug: glargine — 0.3u/kg of glargine, subcutaneously, once
  Arms: Glargine
Drug: saline — 0.3u/kg of saline, subcutaneously, once
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effects of the addition of insulin glargine during the early phase of moderate to severe Diabetic Ketoacidosis (DKA) in children.

The investigators hypothesize that the addition of insulin glargine during the early phase of management of DKA will accelerate acidosis correction, decrease the length of insulin infusion, and decrease the total intensive care unit time in children admitted to the ICU.

ELIGIBILITY:
Inclusion Criteria:

* Ages 6-18 y.o. presenting to Vanderbilt Children's Hospital (VCH) Emergency Room with:
* Established history of insulin dependent diabetes

AND:

* Chief c/o hyperglycemia or vomiting
* Venous pH < 7.24
* Serum Bicarbonate < 18
* Blood glucose > 150
* Urinary Ketones

Exclusion Criteria:

* Age < 6y.o.
* New onset diabetes
* Received IV insulin bolus prior to arrival to VCH Emergency Room (ER)
* Venous pH > 7.24
* Serum Bicarbonate > 18
* Pregnancy
* Received glargine within 12 hours prior to arrival to VCH Emergency Room/Pediatric Critical Care Unit

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 75 (Actual)
Dates: Start 2004-08; Primary Completion 2009-07 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheila McMorrow, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Monroe Carell Children's Hospital, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Original data cannot be found. PI has left Vanderbilt and does not know where records are located. Total enrollment and completion date was obtained from Institutional Review Board records.
Groups:
- Glarine: glargine: 0.3u/kg of glargine, subq, once
- Placebo: saline: 0.3cc/kg of saline, subq, once
Period: Overall Study
Arm/Group | Glarine | Placebo
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Glargine | Placebo | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Time of Acidosis Correction
Description: Unable to find any data on this study. PI left Vanderbilt and there was not a publication.
Time Frame: Minutes
Arm/Group | Glarine | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Time on Insulin Drip
Description: Unable to find any data on this study. PI left Vanderbilt and there was not a publication.
Time Frame: Minutes
Arm/Group | Glarine | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Total Hospital Stay
Description: Unable to find any data on this study. PI left Vanderbilt and there was not a publication.
Time Frame: Days
Arm/Group | Glarine | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Unable to find any data on this study. PI left Vanderbilt and there was not a publication.
Arm/Group | Glarine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No